CLINICAL TRIAL: NCT03226093
Title: Safety Analysis of Implantation of Stromal Vascular Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioheart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-SS-001
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Safety Issues

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stromal Vascular Fraction (Experimental): Isolation of SVF from fat tissue for re-administration into the same patient
  Interventions: Procedure: Stromal Vascular Fraction

INTERVENTIONS:
Procedure: Stromal Vascular Fraction — The fat was separated via centrifuge to isolate the SVF and the cells were delivered intraarticularly, intravenously, intrathecally, or intradiscally directly into the same patient

SUMMARY:
Stromal vascular fraction (SVF) can be isolated from fat (adipose) tissue in an outpatient in-clinic procedure. Platelet rich plasma (PRP) can be isolated from peripheral blood. The SVF includes a variety of different cells and growth factors where the adipocyte (fat cell) population has been removed. The use of SVF in the clinic for a variety of indications is analyzed for incidences of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 97
* Able and willing to give written informed consent
* Up to date on all age and gender appropriate cancer screening

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease patients known to have tested positive for HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis. Will have an expert consulted as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results

Ages: 15 Years to 97 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 12 months
  Collection of adverse events